CLINICAL TRIAL: NCT06406153
Title: A Phase III, Single Arm, Cross-over, Multicenter Clinical Trial to Compare Efficacy and Safety of YW17(Laronidase; CinnaGen) Versus Laronidase (Aldurazyme®; Genzyme, BioMarin) in Patients With Mucopolysaccharidosis Type I (MPS I)"
Brief Title: Efficacy and Safety of YW17 (Laronidase-CinnaGen) Compared to Aldurazyme® in MPS I Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIN.LAR.AR.III.97
Record Dates: First submitted 2024-04-27; First posted 2024-05-09 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Mucopolysaccharidosis Type 1
Keywords: Urinary Glycosaminoglycans; Laronidase; Mucopolysaccharidosis type I; Aldurazyme®
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — Iduronidase; Histamine Antagonists; Antipyretics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YW17 (laronidase biosimilar) (Experimental): YW17 (2.9 mg/5 mL) produced by CinnaGen Company, is administered 0.58 mg/kg weekly.
  Interventions: Biological: Laronidase; Drug: Antihistamine; Drug: Antipyretic
- Aldurazyme® (Active Comparator): Aldurazyme® (2.9 mg/5 mL), is administered 0.58 mg/kg weekly.
  Interventions: Biological: Laronidase; Drug: Antihistamine; Drug: Antipyretic

INTERVENTIONS:
Biological: Laronidase — Laronidase as Aldurazyme® (the first 12 weeks) or YW17 (the second 12 weeks) is administered.
Drug: Antihistamine — An antihistamine is administered one hour before the infusion.
Drug: Antipyretic — An antipyretic is administered one hour before the infusion.

SUMMARY:
The purpose of this phase III study is to assess the efficacy and safety of YW17 produced by CinnaGen Company compared to Aldurazyme® in mucopolysaccharidosis type I (MPS I) patients.

All patients receive Aldurazyme® for 12 weeks, followed by YW17 for another 12 weeks.

The primary outcome is the assessment of the maintenance of the mean uGAG levels at the end of each medication administration. The secondary outcomes are the assessment of 6-minute walking test (6MWT), predicted forced vital capacity (FVC), enzyme activity assay, and adverse events (AEs).

DETAILED DESCRIPTION:
This is a phase III, single-sequence, cross-over study to assess the efficacy and safety of YW17 produced by CinnaGen Company in comparison with Aldurazyme® in MPS I patients.

All patients receive 0.58 mg/kg of Aldurazyme® for 12 weeks and then receive 0.58 mg/kg of YW17 for another 12 weeks.

Premedication with antipyretics and/or antihistamines is administered for all patients one hour before the infusion.

The primary outcome is to compare the mean uGAG levels at weeks 8, 10, and 12 (related to Aldurazyme®) with the mean uGAG levels at weeks 20, 22, and 24 (related to YW17).

The secondary outcomes, including 6MWT and FVC are assessed at the beginning and the end of each medication administration. Enzyme activity is assessed at the end of each medication administration. Safety assessments are performed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-18
* Diagnosed with MPS I
* Signing informed consent form

Exclusion Criteria:

* Prior bone marrow transplantation or being a candidate for receiving haematopoietic stem cell transplantation (HSCT)
* Prior tracheotomy
* Being naïve to laronidase
* Acute hydrocephalus
* Abnormal renal function determined by measuring serum creatinine and blood urea nitrogen (BUN) levels
* Any severe organic disease that is not associated with MPS I
* Known hypersensitivity to laronidase or components of the laronidase solution
* Presence of any medical condition or other circumstances that could significantly interfere with study compliance
* Pregnancy and lactation
* Administration of any investigational drug within 30 days before study enrollment

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
mean uGAG | Baseline, weeks 8, 10, 12, 20, 22, and 24
  urinary glycosaminoglycan

SECONDARY OUTCOMES:
mean 6MWT | Baseline, week 12, week 24
  6-minute walking test
mean predicted FVC | Baseline, week 12, week 24
  Forced vital capacity
mean enzyme activity level | Weeks 11 and 23
  Enzyme activity assay
Number of participants with adverse events | During the study period (screening visit up to week 24)
  All reported AEs are classified based on the Medical Dictionary for Regulatory Activities (MedDRA) terms and are graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rabani, Professor, Principal Investigator — Professor of Pediatric Endocrinology & Metabolism, Department of Pediatrics
Locations (4):
- Iran (4):
  - Clinical Research Development Unit of Akbar Hospital, Faculty of Medicine, Mashhad
  - Growth and Development Research Center, Childrens Medical Center, Tehran
  - Loghman Hospital, Tehran
  - Mofid Childrens Hospital, Tehran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rabbani A, Alaei M, Asl SN, Setoodeh A, Shakiba M, Salehpour S, Eshraghi P, Salehpour O, Sabzvari A, Kafi H, Jarollahi A. Efficacy and safety of a biosimilar laronidase versus the reference laronidase in patients with mucopolysaccharidosis type I. Sci Rep. 2025 Aug 19;15(1):30427. doi: 10.1038/s41598-025-16351-4. PMID 40830667